CLINICAL TRIAL: NCT07376369
Title: Primipar Annelerde Eş Desteğinin Doğum Sonu Ebeveynlik Özgüveni ve Depresyon Düzeyleri Üzerindeki Etkisi: Kesitsel Bir Çalışma
Brief Title: Association of Spousal Support With Parenting Self-Confidence and Depression in Primipar Mothers
Status: Recruiting | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Acibadem University (Other)
Responsible Party: Principal Investigator, Eslem Altıntaş, MSc, Acibadem University
Other Study IDs: 2025-20/738
Record Dates: First submitted 2026-01-22; First posted 2026-01-29 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Support; Postpartum Period; Parenting
Keywords: Postpartum Period; Support; Parenting; Primipar

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primipar mothers: Primipar mothers aged 18 years and older, who are in the postpartum period (0-12 months), living with their spouse/partner, and participating voluntarily in this observational study.

SUMMARY:
The transition to motherhood, particularly for first-time (primiparous) women, is a critical life period requiring substantial psychological and social adjustment. Hormonal changes, increased caregiving responsibilities, sleep disturbances, and potential social isolation during pregnancy and the postpartum period may increase vulnerability to stress, anxiety, and depressive symptoms. Postpartum depression (PPD) is a common mental health concern that adversely affects maternal well-being, mother-infant interaction, and infant development, with insufficient social support identified as one of its most significant risk factors.

Maternal self-efficacy, defined as a mother's perceived competence in caring for and responding to her infant's needs, is a key indicator of successful adaptation to the parenting role. Evidence suggests that maternal self-efficacy develops primarily within the first months after childbirth and tends to be lower in primiparous women. Low parenting self-efficacy has been associated with increased depressive symptoms, higher parenting stress, impaired mother-infant bonding, and negative developmental outcomes for the infant.

Among social support sources, partner support plays a particularly protective role during the transition to parenthood. Emotional, informational, and practical support provided by the partner has been shown to enhance maternal self-efficacy, reduce psychological distress, improve marital adjustment, and lower the risk of postpartum depression. Conversely, low perceived partner support and relationship difficulties are associated with an increased risk of PPD in primiparous mothers.

The aim of this study is to examine the relationship between perceived partner support and postpartum parenting self-efficacy and depressive symptoms in primiparous women. Additionally, the study seeks to evaluate the explanatory and protective role of partner support on maternal self-efficacy and postpartum depression during the early postpartum period.

ELIGIBILITY:
Inclusionsd Criteria:

* Aged 18 years or older
* Primiparous mothers (first childbirth)
* Between 0 and 12 months postpartum
* Living with spouse or partner
* Able to read and write Turkish
* Having access to the internet
* Voluntarily agreeing to participate in the study

Exclusion Criteria:

* Diagnosed neurological disorder
* Diagnosed psychiatric disorder
* Visual impairment preventing completion of questionnaires
* Cognitive impairment preventing completion of questionnaires

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of primiparous mothers aged 18 years and older who are between 0 and 12 months postpartum and living with their spouse or partner. Participants will be recruited online via social media and similar digital platforms and will complete self-report questionnaires.
Sampling Method: Non-Probability Sample
Enrollment: 193 (Estimated)
Dates: Start 2026-01-30 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Introduction Information Forum | At enrollment
  This form was developed by the researchers based on the relevant literature and consists of 29 items designed to assess the sociodemographic, obstetric, and early postpartum experiences of primiparous women. The form includes variables related to partner support, sources of social support, childbirth experience, initiation of breastfeeding, and maternal emotional status. The items were constructed using core variables commonly employed in the assessment of psychosocial status during the postpartum period.
Parenting Self-Confidence (Karitane Parenting Confidence Scale) | At enrollment
  Parenting self-confidence assessed using the Karitane Parenting Confidence Scale (KPCS). The scale consists of 15 items scored on a 4-point Likert scale, with total scores ranging from 0 to 42. Higher scores indicate greater parenting self-confidence.
Perceived Spousal Support measured by the Early Postpartum Perceived Spousal Support Scale | At enrollment
  The Early Postpartum Perceived Spousal Support Scale (ELSKAEDÖ) is a structured self-report questionnaire developed to assess women's perceived spousal support during the early postpartum period. The scale consists of 16 items and includes three subdomains: emotional support (7 items), social support (6 items), and physical support (3 items).
  Items are rated on a 5-point Likert scale. Positively worded items are scored from 1 (strongly disagree) to 5 (strongly agree), while negatively worded items are reverse-coded before calculating the total score.
  The total score ranges from 16 to 80, with higher scores indicating greater perceived spousal support and better psychosocial outcomes, and lower scores indicating insufficient perceived support.
Postpartum Depression (Edinburgh Postnatal Depression Scale) | At enrollment
  Depressive symptoms assessed using the Edinburgh Postnatal Depression Scale (EPDS). The scale includes 10 items scored on a 4-point Likert scale, with total scores ranging from 0 to 30. Higher scores indicate greater risk of postpartum depression.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Coşkun, Ph.D., Principal Investigator — Acibadem University
Locations (1):
- Online study, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Warren, P. L. (2005). First-time mothers: Social support and confidence in infant care. Journal of Advanced Nursing, 50(5), 479-488.
- [Background] Yılmaz, B., & Oskay, Ü. (2021). Karitane Parent Self-Confidence Scale: Turkish validity and reliability study. Cukurova Medical Journal, 46(2), 801-813.